CLINICAL TRIAL: NCT01939652
Title: Restrictive Versus Standard Fluid Regime in Elective Minilaparotomy Abdominal Aortic Aneurysm Repair
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Clinical Center Tuzla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKCTUZLA
Record Dates: First submitted 2013-07-19; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Abdominal Aortic Aneurysm > 5.5 cm Effect of a Restricted Intravenous Fluid Regime on Complications and Hospital Stay After the Minilaparotomy AAA Repair.
Keywords: minilaparotomy; AAA; fluid regime
MeSH Terms: interventions — Colloids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drag: Crystalloids and Colloids (Active Comparator): Drag: Crystalloids and Colloids Intraoperative 10 ml/kg/per hour, postoperative 70-100 ml/per hour
  Interventions: Procedure: Restrictive VS Standard Fluid Regime
- Standard fluid regime (Experimental): Drag: Crystalloids and Colloids Intraoperative 15 ml/kg/per hour, postoperative 150-200 ml/per hour
  Interventions: Drug: Drag: Crystalloids and Colloids

INTERVENTIONS:
Procedure: Restrictive VS Standard Fluid Regime
  Arms: Drag: Crystalloids and Colloids
Drug: Drag: Crystalloids and Colloids
  Arms: Standard fluid regime

SUMMARY:
Elective minilaparatomy abdominal aortic aneurysm (AAA) repair is associated with a significant number of complications involving respiratory, cardiovascular, gastrointestinal and central nervous system, and mortality ranging up to 5%. In our study, we tested the hypothesis that intraoperative and postoperative intravenous restrictive fluid regime reduces postoperative morbidity and mortality and improves the outcome of the treatment of minilaparotomy AAA repair.

DETAILED DESCRIPTION:
We investigate effects of a restricted fluid regime versus standard regimen on complications and hospital stay after minilaparatomy aortic aneurysm repair.

ELIGIBILITY:
Inclusion Criteria:

* AAA more than 5,5 cm in diameter tube graft

Exclusion Criteria:

* emargency comorbidity maligancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of major and minor complications | 30 days

SECONDARY OUTCOMES:
ICU and duration of Hospital stay | 30 days
In-hospital mortality, 30-days mortality | 30 days
Fluid balance (daily and cumulative) | 3 days